CLINICAL TRIAL: NCT01453738
Title: A Randomized, Double Blind, Multicentric, Placebo Controlled, Phase -II Study Assessing the Safety and Efficacy of Intraarticular Ex-vivo Cultured Adult Allogeneic Mesenchymal Stem Cells in Patients With Osteoarthritis of Knee
Brief Title: Allogeneic Mesenchymal Stem Cells in Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stempeutics Research Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRPL/OA/09-10/001
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Osteoarthritis of Knee
Keywords: Osteoarthritis; Knee; Stem cells; Mesenchymal Stem Cells
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ex- vivo cultured adult allogeneic MSCs (Experimental): Single intraarticular dose of allogeneic MSCs suspended in 2-4ml Plasmalyte A followed by 2 ml of Hyaluronan
  Interventions: Biological: Ex- vivo cultured adult allogeneic MSCs
- Plasmalyte-A (Placebo Comparator): Single intraarticular dose of 2ml Plasmalyte
  Interventions: Biological: Plasmalyte-A

INTERVENTIONS:
Biological: Ex- vivo cultured adult allogeneic MSCs — Single intraarticular dose of allogeneic MSCs suspended in 2ml Plasmalyte followed by 2ml of Hyaluronan
  Arms: Ex- vivo cultured adult allogeneic MSCs
Biological: Plasmalyte-A — Single intraarticular dose of 2ml Plasmalyte followed by 2ml Hyaluronan
  Arms: Plasmalyte-A

SUMMARY:
This trial is planed to study if allogeneic mesenchymal stem cells would be safe and beneficial in osteoarthritis of knee joint. This is a double blind study. Different doses of stem cells will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females in the age 40 - 70 years (both inclusive)
2. Radiographic evidence of grade 2 to 3 osteoarthritis based on the Kellgren and Lawrence radiographic criteria.
3. History of primary idiopathic osteoarthritis of the knee characterized by pain which requires intake of analgesics.
4. Self-reported difficulty in at least one of the following activities attributed to knee pain: lifting and carrying groceries, walking 400 metres, getting in and out of a chair, or going up and down stairs.
5. Patients who have been on stable medication which may be NSAIDs / Opioid or opiate analgesics, for the past three months.
6. Female patients of childbearing age must be willing to use accepted methods of contraception during the course of the study
7. Ability to provide written informed consent.

Exclusion Criteria:

1. Prior or ongoing medical conditions (e.g., concomitant illness, psychiatric condition, alcoholism, drug abuse), medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.
2. History of surgery, or major trauma to the study joint
3. Arthroscopy on the study joint in the previous 12 months
4. Signs of active study joint inflammation including redness, warmth, and/or, if qualifying with osteoarthritis of the knee, a large, bulging effusion of the study knee joint with the loss of normal contour of the joint at the screening visit or at the baseline examination
5. Patients who had received intraarticular steroids or hyaluronan within the last three months.
6. Infections in or around the knee.
7. Patients awaiting a replacement knee or hip joint
8. Patients with other conditions that cause pain
9. Patients with deformity of the knee joint.
10. Significantly incapacitated or disabled and would be categorized as ACR Functional Class IV (largely or wholly incapacitated), or unable to walk without assistive devices
11. Patients with other known rheumatic or inflammatory disease such as rheumatoid arthritis
12. Other pathologic lesions on x-rays of knee
13. Positive hepatitis B surface antigen, hepatitis C antibody test, Anti human immunodeficiency virus (HIV) antibody test, or RPR
14. History of Bleeding disorders
15. Known hypersensitivity to Hyaluronan products or animal sera
16. For women of child-bearing potential: positive pregnancy test or lactating [Females who are planning pregnancy within next one year should be excluded]

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients with adverse events as a measure of safety and tolerability | 2 years
  * Safety evaluation will include assessment of physical examination, periodic monitoring of vital signs (heart rate, respiratory rate, blood pressure and temperature), clinical laboratory investigations (including haematology, serum chemistry, LFT, urine-analysis) and 12-lead ECG recording.
  * Tolerability: Adverse events monitored using information volunteered by the patients and as observed by the PI will be summarized descriptively by total number of AE(s) and compared between the study arms.

SECONDARY OUTCOMES:
Change from baseline in the WOMAC OA (Western Ontario and McMaster Universities Osteoarthritis) Index -pain subscale score | 2 years
Change from baseline in WOMAC OA stiffness index | 2 years
Change from baseline in WOMAC OA composite index | 2 years
Change from baseline in ICOAP (Intermittent and Constant Osteoarthritis Pain) | 2 years
Change from baseline in radiographic (X-ray) findings of knee | 2 years
Change from baseline in the WORMS score (Whole-Organ Magnetic Resonance Imaging Score) of knee using MRI | 2 years
Change from baseline in arthritis pain scores on the visual analogue scale | 2 years
Reduction in the intake of analgesic tablets from baseline | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Agarwal, MD., DM, Principal Investigator — Department of Immunology Sanjay Gandhi Post Graduate Institute of Medical Sciences; Vivek Pandey, MS, Principal Investigator — Department of Orthopedics, Kasturba Medical College; Naresh Shetty, MS, Principal Investigator — Department of Orthopedics, M. S. Ramaiah Memorial Hospital; Shrikant Wagh, MD, Principal Investigator — Jehangir Hospital; Bhibas Dasgupta, MS, Principal Investigator — Seth G. S. Medical College and KEM Hospital
Locations (5):
- India (5):
  - Department of Orthopedics, M. S. Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Department of Orthopedics, Kasturba Medical College, Manipal, Karnataka
  - Seth G. S. Medical College and KEM Hospital, Mumbai, Maharashtra
  - Jehangir Hospital, Pune, Maharashtra
  - Department of Immunology Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow, Uttar Pradesh

REFERENCES:
- [Derived] Gupta PK, Chullikana A, Rengasamy M, Shetty N, Pandey V, Agarwal V, Wagh SY, Vellotare PK, Damodaran D, Viswanathan P, Thej C, Balasubramanian S, Majumdar AS. Efficacy and safety of adult human bone marrow-derived, cultured, pooled, allogeneic mesenchymal stromal cells (Stempeucel(R)): preclinical and clinical trial in osteoarthritis of the knee joint. Arthritis Res Ther. 2016 Dec 20;18(1):301. doi: 10.1186/s13075-016-1195-7. PMID 27993154